CLINICAL TRIAL: NCT00876291
Title: The Use of Lactobacillus gg in Functional Abdominal Pain in Children: a Double-blind Randomized Control Trial
Brief Title: Efficacy of Lactobacillus GG (LGG) in Children With Abdominal Pain
Acronym: LGGDAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Collaborators: Clinica PEdiatrica Ospedale San Paolo Bari Italy (Unknown)
Responsible Party: Clinica Pediatrica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UB2712
Record Dates: First submitted 2009-04-02; First posted 2009-04-06 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2009-04

CONDITIONS: Functional Abdominal Pain
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo which consisted of capsules identical in taste and appearance to the active study product except for the absence of freeze-dried LGG (and cryoprotectants)
  Interventions: Dietary Supplement: Placebo
- Probiotic (Active Comparator): LGG capsules: each cp containing 3 × 109 colony forming units, CFU
  Interventions: Dietary Supplement: Lactobacillus GG (probiotic )

INTERVENTIONS:
Dietary Supplement: Lactobacillus GG (probiotic ) — LGG capsules: each cp containing 3 × 109 colony forming units, CFU
  Arms: Probiotic
Dietary Supplement: Placebo — placebo which consisted of capsules identical in taste and appearance to the active study product except for the absence of freeze-dried LGG (and cryoprotectants)
  Arms: Placebo

SUMMARY:
Probiotics play an important role in preventing overgrowth of potentially pathogenic bacteria and maintaining the integrity of the gut mucosal barrier. The beneficial effects of probiotics have been previously studied in adult patients with IBS. Even though most of the studies demonstrate efficacy, other studies do not support these observations. Few studies addresses the efficacy of probiotics in children with IBS. The goal of the present study was to determine whether oral administration of the probiotic Lactobacillus GG under randomized, double-blind, placebo-controlled conditions would improve symptoms of children with abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients were considered for study inclusion, if they were 4 - 12 years of age and had if they had a pain history of at least 12 weeks (which need not be consecutive) in the preceding 12 months suggestive for IBS or FAP with no structural or metabolic abnormalities to explain the symptoms and according to the Rome II diagnostic criteria valid at the time of the design of the study.
* IBS was diagnosed in presence of an abdominal discomfort or pain with at least two of three features:

  * relieved with defecation
  * onset associated with a change in stool frequency
  * onset associated with a change in the form (appearance) of the stool.
* FAP was diagnosed in presence of symptoms of
* Continuous (nearly continuous) abdominal pain
* No or only occasional relation of pain with physiological events (e.g. eating, menses)
* Some loss of daily functioning
* The pain is not feigned (e.g. malingering)
* The patient has insufficient criteria for other functional gastrointestinal disorders that would explain the abdominal pain.

Exclusion Criteria:

* Known concomitant psychiatric, neurological, metabolic, hepatic, renal, infectious, haematological, cardiovascular and pulmonary disease
* Treatment with antibiotics/probiotics in the last 2 months
* A pain history suggestive for functional dyspepsia or aerophagia or abdominal migrain
* Growth failure
* Gastroparesis
* Gastrointestinal obstructions/stricture
* Any disease that may affect bowel motility such as diabetes, connective disease or poorly controlled hypo/hyperthyrodism
* Previous abdominal surgery.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2004-12; Primary Completion 2007-12 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was defined as reduction of pain (both number of episodes and intensity) at the end of the intervention. | 12 weeks and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruggiero Francavilla, MD PhD, Principal Investigator — University of Bari
Locations (1):
- Clinica Pediatrica, Bari, Italy

REFERENCES:
- [Derived] Francavilla R, Miniello V, Magista AM, De Canio A, Bucci N, Gagliardi F, Lionetti E, Castellaneta S, Polimeno L, Peccarisi L, Indrio F, Cavallo L. A randomized controlled trial of Lactobacillus GG in children with functional abdominal pain. Pediatrics. 2010 Dec;126(6):e1445-52. doi: 10.1542/peds.2010-0467. Epub 2010 Nov 15. PMID 21078735